CLINICAL TRIAL: NCT04784949
Title: Outcome of PRF Pulpotomy Using Different Bioceramic Materials in Permanent Molars With Irreversible Pulpitis: A Randomized Controlled Trial
Brief Title: PRF Pulpotomy Using Different Bioceramic Materials in Permanent Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mohamed Nageh, Lecturer of Endodontics, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRF Pulp
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Irreversible Pulpitis
Keywords: PRF; Vital pulp therapy; pulpotomy; bioceramics
MeSH Terms: interventions — Dental Cements; mineral trioxide aggregate; tricalcium silicate

STUDY DESIGN:
Intervention Model Description: permanent molar with symptomatic irreversible pulpitis
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Portland cement (Experimental): pulpotomy with PRF and white Portland cement
  Interventions: Procedure: portland cement
- Mineral trioxide aggregate (Experimental): pulpotomy with PRF and Mineral trioxide aggregate
  Interventions: Procedure: Mineral trioxide aggregate
- Biodentine (Experimental): pulpotomy with PRF and Biodentine
  Interventions: Procedure: Biodentine

INTERVENTIONS:
Procedure: portland cement — pulpotomy with PRF and white Portland cement
  Arms: Portland cement
Procedure: Mineral trioxide aggregate — pulpotomy with PRF and white Mineral trioxide aggregate
  Arms: Mineral trioxide aggregate
Procedure: Biodentine — pulpotomy with PRF and Biodentine
  Arms: Biodentine

SUMMARY:
this study aimed to compare the clinical and radiographic outcomes of full pulpotmy after application of Biodentine, or MTA, or Portland cement above PRF membrane In permanent molars with irreversible pulpitis

ELIGIBILITY:
Inclusion Criteria:

* spontaneous, lingering pain exacerbated by hot and cold , and/or radiating pain
* Responded to cold and electric pulp testing

Exclusion Criteria:

* pain on palpation, percussion,
* mobility or swelling
* peridontall widening
* Teeth with marginal periodontitis or crestal bone loss
* resorption
* calcified canals

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Change in postoperative pain | 24 hours, 48 hours, 1 week, every 3 months for 12 months
  persistence , relief , or exacerbation of pain using visual analogue scale for pain score
Change in swelling | 24 hours, 48 hours, 1 week, every 3 months for 12 months
  appearance of periapical swelling or facial swelling after the clinical procedures (Binary outcome: Yes/No)
Change in Mobility | 24 hours, 48 hours, 1 week, every 3 months for 12 months
  appearance of teeth mobility after the clinical procedures (record of periodontal pocket depth)

SECONDARY OUTCOMES:
calcific like bridge | 12 month
  measure of the calcific bridge thickness using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asgary S, Eghbal MJ. Treatment outcomes of pulpotomy in permanent molars with irreversible pulpitis using biomaterials: a multi-center randomized controlled trial. Acta Odontol Scand. 2013 Jan;71(1):130-6. doi: 10.3109/00016357.2011.654251. Epub 2012 Feb 20. PMID 22339289
- [Background] Cushley S, Duncan HF, Lappin MJ, Tomson PL, Lundy FT, Cooper P, Clarke M, El Karim IA. Pulpotomy for mature carious teeth with symptoms of irreversible pulpitis: A systematic review. J Dent. 2019 Sep;88:103158. doi: 10.1016/j.jdent.2019.06.005. Epub 2019 Jun 20. PMID 31229496